CLINICAL TRIAL: NCT00943787
Title: Counter-regulatory Impairment and the Effect of Microvascular Insulin Transfer in Type 1 Diabetes Mellitus
Acronym: BPK003
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Boris Kovatchev, PhD, Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 12252
Record Dates: First submitted 2009-06-24; First posted 2009-07-22 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (1):
- SMBG followed by clamp (Other): One month of self-monitored blood glucose (SMBG) field data was used to calculate measures of glucose variability and risk of hypoglycemia, while the hyperinsulinemic, euglycemic and hypoglycemic clamp procedure was used to evaluate insulin sensitivity and epinephrine response during induced hypoglycemia.
  Interventions: Procedure: Hyperinsulinemic, euglycemic and hypoglycemic clamp

INTERVENTIONS:
Procedure: Hyperinsulinemic, euglycemic and hypoglycemic clamp — At 21:30h, an overnight insulin infusion was titrated to control the subjects' BG overnight between 100 and 150mg/dL by blood sampling for plasma glucose via a YSI analyzer every 30min and adjusting the rate of insulin infusion as needed. At the beginning of the clamp, the overnight insulin was replaced by an insulin infusion via a Harvard pump given as a 20mU/kg priming over a 10-min period, followed by a constant rate delivery of 1mU/kg/min until the end of the clamp. Blood was sampled for plasma glucose, and glucose was clamped at basal levels for the euglycemic control period of 150min via a variable-rate infusion of 20% dextrose. Then the glucose concentration was lowered at a rate of 1mg/dL/min to a minimum of 50mg/dL, where it was held constant for 30min. Finally, the glucose concentration was increased at a rate of 1mg/dL/min to 90mg/dL, where it was held for an additional 30min. Blood was sampled for epinephrine during euglycemia, hypoglycemia, and recovery.

SUMMARY:
The researchers plan to test the following hypothesis:

A good level of glucose control in Type 1 Diabetes Mellitus (T1DM) is dependent on two levels of feedback from the body:

1. the transport of insulin through small blood vessels: suggesting that hypoglycemia leads to increased insulin sensitivity which then causes recurrent hypoglycemia;
2. the endocrine level, defined as insulin-glucose interaction and hormonal counter-regulation.

The researchers plan to investigate the relationships between hypoglycemia, insulin transport, and counter-regulation. This study will ultimately lead to a better understanding of risk for recurrent hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Participated in and satisfied all of the inclusion criteria of NCT00315939
* 18 years of age or older
* Have Type 1 Diabetes Mellitus defined by American Diabetes Association criteria or judgment of physician
* Since our major goal is the investigation of hypoglycemia, we will preferentially recruit patients with a history of severe hypoglycemia/moderate hypoglycemia anticipating that approximately (~) half of the recruited subjects will have had two or more severe or moderate hypoglycemia episodes in the past 12 months

Exclusion Criteria:

* Age < 18
* Pregnancy
* Use of oral steroids
* Hematocrit < 36% (females); < 38% (males)
* Symptomatic heart disease (e.g., history of myocardial infarction, history of coronary bypass or stenting procedure, angina, episode of chest pain of cardiac etiology with documented EKG changes, positive stress test or catheterization with coronary blockages > 50%)
* History of an ischemic cerebrovascular event
* Active substance abuse
* Psychosis
* Mental retardation
* Severe depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Kovatchev, Ph.D., Principal Investigator — University of Virginia Health Systems - Behavioral Medicine Center
Locations (1):
- University of Virginia Health System - Behavioral Medicine Center, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Pitsillides AN, Anderson SM, Kovatchev B. Hypoglycemia risk and glucose variability indices derived from routine self-monitoring of blood glucose are related to laboratory measures of insulin sensitivity and epinephrine counterregulation. Diabetes Technol Ther. 2011 Jan;13(1):11-7. doi: 10.1089/dia.2010.0103. PMID 21175266
- [Derived] Chan A, Barrett EJ, Anderson SM, Kovatchev BP, Breton MD. Muscle microvascular recruitment predicts insulin sensitivity in middle-aged patients with type 1 diabetes mellitus. Diabetologia. 2012 Mar;55(3):729-36. doi: 10.1007/s00125-011-2402-3. Epub 2011 Dec 14. PMID 22167126

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 2/2006-5/2009. Recruitment included outpatients at UVA clinics, former research subjects, and local advertising. All subjects ≥18 years of age and had type 1 diabetes defined by American Diabetes Association criteria or judgment of the study endocrinologist after review of the clinical history.
Groups:
- Adults With T1DM From Subjects: Subjects with type 1 diabetes performed self-monitoring of blood glucose (SMBG) for a month, followed by an inpatient hyperinsulinemic euglycemic and hypoglycemic clamp. SMBG field data were used to calculate measures of glucose variability and risk of hypoglycemia, while the clamp procedure was used to evaluate insulin sensitivity and epinephrine response during induced hypoglycemia.
Period: Overall Study
Arm/Group | Adults With T1DM From Subjects
Started | 41
Completed | 34
Not Completed | 7
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Adults With T1DM From Subjects
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 34
Glycosylated hembglobin (HbA1c) [Mean (Standard Deviation); unit: percent] | 7.6 (0.21)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Epinephrine Response (LBGI Groups)
Description: Mean maximum epinephrine response during induced hypoglycemia is the average of subjects' maximum concentration of all epinephrine measurements taken at plasma glucose level lower than 70mg/dL.
  Low blood glucose index (LBGI) is a metric to calculate the risk for hypoglycemia based on frequency and extent of past events based on SMBG readings. In studies, the LBGI typically accounted for 40-55% of the variance of future significant hypoglycemia in the subsequent 3-6 months. The LBGI has established risk categories: Low Risk, LBGI < 2.5; Moderate Risk, 2.5 < LBGI < 5; and High Risk, LBGI > 5, indicating an over 10-fold increase in future severe hypoglycemia from the lowest to the highest risk category.
Time Frame: 285 min (time of clamp)
Population: 3 participants did not have adequate epinephrine data.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Adults With T1DM From Subjects
Number analyzed (Participants) | 31
pg/ml
  LBGI < 2.5 | 495 (60)
  LBGI >= 2.5 | 217 (40)

2. Secondary Outcome: Maximum Epinephrine Response (ADRR Groups)
Description: Mean maximum epinephrine response during induced hypoglycemia is the average of subjects' maximum concentration of all epinephrine measurements taken at plasma glucose level lower than 70mg/dL.
  Average Daily Risk Range (ADRR) is associated with glycemic variability and risk of both hyper- and hypoglycemia.
  Low Risk, ADRR < 20; Moderate Risk, 20 < ADRR < 40; and High Risk,ADRR > 40.
Time Frame: 285 min (time of clamp)
Population: 3 participants did not have enough epinephrine data
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Adults With T1DM From Subjects
Number analyzed (Participants) | 31
pg/ml
  ADRR < 40 | 417 (45)
  ADRR >= 40 | 167 (45)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Adults With T1DM From Subjects
Serious Adverse Events (participants affected / at risk) | 3/34
Other Adverse Events (participants affected / at risk) | 8/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults With T1DM From Subjects (N=34)
Orthostatic Hypotension (Vascular disorders) | 2 (2)
Vasovagal Hypotension (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults With T1DM From Subjects (N=34)
Hyperglycemia (Endocrine disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Lower Back Pain (General disorders) | 1 (1)
Abdomen ecchymosis near Guardian site (Skin and subcutaneous tissue disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes